CLINICAL TRIAL: NCT01107509
Title: A Pilot Study of Neo-Adjuvant Everolimus in Patients With Advanced Renal Cell Carcinoma Undergoing Definitive Therapy With Radical Nephrectomy, or Cytoreductive Nephrectomy - Analysis of Serum and Tissue Biomarkers
Brief Title: Pilot Study of Neo-Adjuvant Everolimus to Treat Advanced Renal Cell Carcinoma - Analysis of Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIURCCEVERO
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal cell carcinoma; Metastatic; everolimus; neo-adjuvant; biomarkers; nephrectomy; Locally advanced clear cell renal carcinoma; Metastatic clear cell renal carcinoma; Clear Cell Renal Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neo-adjuvant everolimus (Experimental)
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — 10 mg/ day everolimus in the form of an oral tablet for 12 weeks leading up to nephrectomy (with a 1-week perioperative washout period) in patients with locally advanced disease and re-initiating the drug postoperatively in patients with metastatic disease for up to 24 months, or until disease progression. Dosage may be reduced at any point to 5 mg/ day in the event of any grade 3/ 4 toxicity.
  Other Names: Afinitor; RAD-001

SUMMARY:
This study will gather data on potential biomarkers in the treatment of advanced renal cell carcinoma (kidney cancer) and investigate their use as indicators of disease response. The results could eventually enable doctors to match levels of therapy to levels of biomarker on an individual basis and to increase the chance of disease response in patients. This study will also test a new paradigm in the treatment approach of advanced kidney cancer by using the drug everolimus in a neo-adjuvant setting, with the overarching goal of decreasing cancer recurrence rates and improving patient outcomes and survival.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and capable of giving informed consent
* Radiological evidence of RCC consisting of: CT scan with stage T2, T3, T3a, T3b, T4, or any stage T with N1/ 2 and/ or metastatic disease
* Having a nephrectomy and willing to have a kidney biopsy
* ECOG score 0 or 1
* Clear cell histology
* Negative for HIV, Hepatitis B, and Hepatitis C
* Negative pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Stage T1 disease without metastases
* Abnormal laboratory values at screening within the following ranges:
* Absolute neutrophil count ≤ 1.5 × 109/ L; Platelet count ≤ 100 × 109/ L
* Leukocyte count ≤ 3 × 109/ L; Hemoglobin ≤ 80 g/ L; Serum creatinine ≥ 2.0 × the upper normal limit (UNL); Total bilirubin ≤ 1.5 × UNL; AST and ALT ≤ 3.0 × UNL
* Fasting serum cholesterol ≤ 9.0 mmol/ L; Fasting serum triglycerides ≥ 5.0 mmol/L
* Any major illness that, based on the investigator's judgment, will substantially increase the risk associated with a subject's participation in this study
* Other currently active malignancies
* Currently taking any medications known to interfere with the metabolism of everolimus
* Receiving anticoagulation with warfarin
* A history of pulmonary hypertension or interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Response of primary tumor and metastases (if applicable) to everolimus in terms of tumor size and appearance (RECIST imaging response criteria) as determined by CT or MRI | From 6 weeks after starting neo-adjuvant everolimus until 1 year post-nephrectomy (or up to 24 months post-nephrectomy in metastatic patients)

SECONDARY OUTCOMES:
Effect of everolimus on blood and tissue biomarker expression (periodic blood testing and tissue samples from baseline renal biopsy and nephrectomy) in and among patients with locally advanced and metastatic disease with respect to baseline values | From baseline to 1 year post-nephrectomy for blood biomarker levels and from baseline to nephrectomy (week 12) for tissue biomarker levels

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada